CLINICAL TRIAL: NCT01029314
Title: Pilot Study of the Genius(TM)2 Tympanic Thermometer in Cardiac Patients Requiring Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Tyco Healthcare Group (Industry)
Responsible Party: Edwin Avery IV, MD, Principal Investigator, Massachusetts General Hospital Corporation
Other Study IDs: 353.29
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Cardiac Surgical Procedures
Keywords: Thermometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiopulmonary bypass surgery: Thirty to fifty cardiac surgery patients undergoing cardiopulmonary bypass will have serial triplicate temperatures taken by both the Genius 2 tympanic thermometer and the Exergen-TAT 5000 temporal artery thermometer at predetermined perioperative time points. These temperature readings will be compared to at least one core temperature (i.e., pulmonary artery).

SUMMARY:
Primary study objective is to test the accuracy of the Genius 2 tympanic thermometer and the Exergen TAT-5000(TM) temporal artery thermometer as compared with serial perioperative core temperature measurements obtained in cardiac surgical patients during cardiopulmonary bypass. Study hypothesis: The Genius 2 thermometer will display greater precision and accuracy than the Exergen TAT-5000 thermometer when compared to core body temperature in patients undergoing CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult subjects greater than/equal to 18 years of age providing signed informed consent
* Febrile or afebrile
* Planned monitoring of core temperature at a minimum of two separate sites, one of which includes the pulmonary artery
* Planned use of cardiopulmonary bypass for a cardiac surgical procedure.

Exclusion Criteria:

* Mist tents or oxygen hoods
* Hot or cold applications to the head
* Patients that have the planned use of deep hypothermic circulatory arrest
* Aural anomalies (e.g., external auditory canal less than 2cm in length, persistent ear pain)
* Any other major anomaly, surgery or medical condition precluding participation according to manufacturers' stated exclusions or in the opinion of the principal investigator
* Blood, cerumen, excessive hair, inflammation, infection, ulceration or foreign object in the ear observed by otoscopic examination
* Any other signs or symptoms of distress or a condition which would, or in the opinion of the principal investigator, render their participation in the study detrimental to their well-being.
* Previous refusal or enrollment in this study
* Previous or concurrent participation in a clinical trial of a drug or device within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults greater than/equal to 18 years of age scheduled for a cardiac surgical procedure requiring cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Thermometer accuracy and precision: 1) Temperature obtained by Genius 2 and Exergen compared to core body temperature (accuracy). 2) Agreement among temperatures taken in triplicate at a given time point (precision). | Subjects are followed for temperature collection until 6 hours post admission to the intensive care unit; lab data and patient outcomes are collected until the time of hospital discharge.

SECONDARY OUTCOMES:
Effect of environmental conditions before, during and after surgery, on body temperature and thermometer performance (ambient temperature, humidity, diaphoresis, warming devices). | Predetermined perioperative time periods up to 6 hours after intensive care unit admission.
Explore possible relationships between temperature management and duration of CABG surgery and the following patient outcomes: mortality, renal failure (new onset), stroke, myocardial infarction, length of hospital stay, length of ICU stay. | Predetermined perioperative time periods until hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Avery, MD, Principal Investigator — Massachusetts General Hospital Corporation
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States